CLINICAL TRIAL: NCT04531046
Title: Phase 2, Open-Label Study Evaluating Axi-Cel as a 2nd Line Therapy in Patients With Relapsed/Refractory Aggressive B-Non Hodgkin Lymphoma (B-NHL) Who Are Ineligible to Autologous Stem Cell Transplantation
Brief Title: Axi-Cel as a 2nd Line Therapy in Patients With Relapsed/Refractory Aggressive B Lymphoma Ineligible to Autologous Stem Cell Transplantation
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Lymphoma Academic Research Organisation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALYCANTE
Record Dates: First submitted 2020-08-25; First posted 2020-08-28 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: B-Cell Lymphoma Refractory; B-cell Lymphoma Recurrent
MeSH Terms: interventions — axicabtagene ciloleucel

STUDY DESIGN:
Intervention Model Description: open-label, multicenter study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- axicabtagene ciloleucel (Experimental): Single infusion administered intravenously at a target dose of 2 x 10^6 anti-CD19 CAR T cells/kg
  Interventions: Drug: axicabtagene ciloleucel

INTERVENTIONS:
Drug: axicabtagene ciloleucel — Patient-specific (autologous) product cryopreserved in cryostorage bag
  Other Names: axi-cel

SUMMARY:
This is a phase 2, open-label, multicenter study evaluating axicabtagene ciloleucel (axi-cel) as a 2nd line therapy in patients with Relapsed/Refractory aggressive B-NHL who are ineligible to receive Autologous Stem Cell Transplantation but eligible to receive CAR T-cell therapy.

DETAILED DESCRIPTION:
Axicabtagene ciloleucel (axi-cel) is a chimeric antigen receptor (CAR) T-cell therapy directed against CD19 which has been approved for the treatment of relapse/refractory diffuse large B-cell lymphoma DLBCL and primary mediastinal large B-cell lymphoma (PMBCL) after 2 or more lines of systemic therapy.

But administrating CAR T-cells earlier in the therapeutic strategy may be beneficial to patients.

Axi-cel will improve the outcome of patients with DLBCL who are refractory or relapse early (i.e. within 1 year from end of treatment) after first-line therapy and who are not eligible for Autologous Stem Cell Transplantation (ASCT).

Transplant-ineligible patients will include those who are deemed ineligible for high-dose chemotherapy and Hematopoietic Stem Cell Transplantation (HSCT) due to age, comorbidity, or prior ASCT.

The primary endpoint will be complete metabolic response (CMR) at 3 months after Axi-cel infusion.

ELIGIBILITY:
Inclusion Criteria:

* Patient who understands and speaks one of the country official languages and signed Informed Consent Form
* Histologically proven relapsed or refractory aggressive B-cell non-Hodgkin lymphoma (B-NHL) of the following histology at relapse: diffuse large B-cell lymphoma (DLBCL), high-grade B-cell lymphoma (HGBL), follicular lymphoma Grade 3B per World Health Organization (WHO) 2016 classification and Primary mediastinal Bcell lymphomas. Indolent B-NHL who transformed into aggressive B-NHL and were previously treated with Rituximab-Cyclophosphamide, Hydroxydaunomycin, Oncovin, and Prednisone (R-CHOP) are eligible.
* Tumoral tissue (at diagnosis or relapse) available for central pathology review, exploratory endpoints and ancillary studies
* Positron-emission tomography (PET)-positive disease
* Patients must have received adequate first-line therapy including at a minimum: an anti-CD20 monoclonal antibody (rituximab or obinutuzumab), and Cyclophosphamide, Hydroxydaunomycin, Oncovin, and Prednisone (CHOP) or CHOP-like chemotherapy
* Relapsed or refractory disease after first-line chemoimmunotherapy (full dose of R-CHOP or R-CHOP-like regimen), documented by PET-scan
* At least 2 weeks must have elapsed since any prior systemic cancer therapy at the time the patient provides consent
* Patients must be autologous stem cell transplantation (ASCT)-ineligible
* Patients must be CAR-T-eligible
* Females of childbearing potential must have a negative serum or urine pregnancy test (females who have undergone surgical sterilization or who have been postmenopausal for at least 12 months are not considered to be of childbearing potential)

Exclusion Criteria:

* Patients who received more than one prior line of systemic therapy
* Patients who are intolerant to first-line therapy or who received suboptimal first-line therapy, including dose-reduced R-CHOP ("R-miniCHOP"), and those who discontinued prematurely first-line therapy due to toxicity are not eligible
* Prior CD19 targeted therapy
* Patients with cardiac atrial or cardiac ventricular lymphoma involvement
* Requirement for urgent therapy due to tumor mass effects, such as bowel obstruction or blood vessel compression
* Patient with clinically significant pleural effusion
* History of another primary malignancy that has not been in remission for at least 2 years (except for nonmelanoma skin cancer or carcinoma in situ (eg, cervix, bladder, breast))
* Patients with detectable Central Nervous System (CNS) lymphoma
* History or presence of non-malignant CNS disorder, such as seizure disorder requiring anti-convulsive therapy, cerebellar disease, or any autoimmune disease with CNS involvement disease
* Active hepatitis B or hepatitis C infection, positive serology of human immunodeficiency virus (HIV) and syphilis at the time of screening
* Uncontrolled systemic fungal, bacterial, viral or other infection despite appropriate antibiotics or other treatment at the time of leukapheresis or axi-cel administration
* History of any one of the following cardiovascular conditions within the past 6 months: Class III or IV heart failure as defined by the New York Heart Association, cardiac angioplasty or stenting, myocardial infarction, unstable angina, or other clinically significant cardiac disease
* History of autoimmune disease requiring systemic immunosuppression and/or systemic disease modifying agents within the last year
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis per chest computed tomography (CT) scan at screening.
* History of severe immediate hypersensitivity reaction to tocilizumab or any of the agents used in this study
* History of severe immediate hypersensitivity reaction attributed to aminoglycosides, cyclophosphamide and fludarabine
* Treatment with a live, attenuated vaccine within 6 weeks prior to initiation of study treatment or anticipation of need for such a vaccine during the course of the study
* Women of childbearing potential who are pregnant or breastfeeding (from the time of consent during treatment and for at least 6 months after conditioning chemotherapy dosing or axicabtagene ciloleucel dosing, whichever is later)
* In the investigator's judgment, the patient is unlikely to complete all protocol-required study visits or procedures, including follow-up visits, or comply with the study requirements for participation
* Adult person unable to provide informed consent because of intellectual impairment, any serious medical condition, laboratory abnormality or psychiatric illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2022-04-19 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Complete Metabolic Response (CMR) - determined by investigator | 3 months from axi-cel infusion
  CMR from axi-cel infusion (without additional anticancer therapy) based on investigator disease assessment according to PET-scan (using the Lugano Response Criteria)

SECONDARY OUTCOMES:
Complete Metabolic Response (CMR) - determined by central imaging review | 3 months from axi-cel infusion
  CMR from axi-cel infusion (without additional anticancer therapy) determined by central imaging review (using the Lugano Response Criteria)
Best objective response | between Day 14 and Month 12
  Percentage of CMR and Partial MR determined by investigator disease assessment
Number of Serious Adverse Events (SAE) | at 30 days after axi-cel infusion
Event-free survival (EFS) based on investigator disease assessment | at 3 months
Event-free survival (EFS) based on investigator disease assessment | at 6 months
Event-free survival (EFS) based on investigator disease assessment | at 12 months
Event-free survival (EFS) based on central imaging review | at 3 months
Event-free survival (EFS) based on central imaging review | at 6 months
Event-free survival (EFS) based on central imaging review | at 12 months
Modified EFS (mEFS) based on investigator assessment | at 6 months
Modified EFS (mEFS) based on investigator assessment | at 12 months
Modified EFS (mEFS) based on central imaging review | at 6 months
Modified EFS (mEFS) based on central imaging review | at 12 months
Best objective response | at 2 years
Best objective response | at 3 years
Duration of response (DOR) | at 2 years
Duration of response (DOR) | at 3 years
Overall survival (OS) from leukaphaeresis and Axi-cel infusion | at 2 years
Overall survival (OS) from leukaphaeresis and Axi-cel infusion | at 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Roch Houot, PhD, Principal Investigator — Rennes University Hospital, Rennes, France; François Lemonnier, PhD, Principal Investigator — Henri Mondor Hospital, Créteil, France
Locations (16):
- CH Liège, Liège, Belgium
- France (15):
  - CHU de Bordeaux - Hôpital Haut Lévêque, Bordeaux
  - CHU Clermont Ferrand - Hôpital Estaing, Clermont-Ferrand
  - APHP - Hôpital Henri Mondor, Créteil
  - CHU de Dijon - Hôpital le Bocage, Dijon
  - Hôpital Claude Huriez, Lille
  - Hôpital Saint Eloi, Montpellier
  - CHU de Nantes - Hôtel Dieu, Nantes
  - APHP - Hôpital Saint Louis, Paris
  - Hopital La Pitié Salpétriere, Paris
  - Hôpital Saint Antoine, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU de Rennes - Hôpital de Pontchaillou, Rennes
  - IUCT Oncopole, Toulouse
  - CHU Brabois, Vandœuvre-lès-Nancy
  - Institut de Cancérologie Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Charton E, Anota A, Bachy E, Cartron G, Gros FX, Morschhauser F, Oberic L, Gastinne T, Feugier P, Dulery R, Thieblemont C, Joris M, Jardin F, Choquet S, Casasnovas RO, Brisou G, Cheminant M, Bay JO, Llamas Gutierrez F, Portugues C, Itti E, Palard-Novello X, Blanc-Durand P, Al Tabaa Y, Bailly C, Laurent C, Lemonnier F, Houot R. Health-related quality of life after second-line Axi-cel in transplant-ineligible patients with large B-cell lymphoma. Blood Adv. 2026 Jan 9:bloodadvances.2025018057. doi: 10.1182/bloodadvances.2025018057. Online ahead of print. PMID 41512176
- [Derived] Houot R, Bachy E, Cartron G, Gros FX, Morschhauser F, Oberic L, Gastinne T, Feugier P, Dulery R, Thieblemont C, Joris M, Jardin F, Choquet S, Casasnovas O, Brisou G, Cheminant M, Bay JO, Gutierrez FL, Menard C, Tarte K, Delfau MH, Portugues C, Itti E, Palard-Novello X, Blanc-Durand P, Al Tabaa Y, Bailly C, Laurent C, Lemonnier F. Axicabtagene ciloleucel as second-line therapy in large B cell lymphoma ineligible for autologous stem cell transplantation: a phase 2 trial. Nat Med. 2023 Oct;29(10):2593-2601. doi: 10.1038/s41591-023-02572-5. Epub 2023 Sep 14. PMID 37710005